CLINICAL TRIAL: NCT04820101
Title: Dexmedetomidine for LISA Procedure in Preterm Infants: a Pilot Study
Brief Title: Dexmedetomidine for LISA Procedure in Preterm Infants
Acronym: DEXLISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Paola Lago, Head of Neonatal Intensive Care Unit, Principal Investigator, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEXLISA 920/CE Marca
Record Dates: First submitted 2021-03-19; First posted 2021-03-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: RDS
Keywords: RDS; LISA; preterm; sedation; dexmedetomidine
MeSH Terms: conditions — Premature Birth | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Every preterm newborns 26+0 -36+6 wGA with RDS needing surfactant therapy (Experimental): Every preterm newborns 26+0-36+6 wGA who undergoes LISA procedure will receive sedation with dexmedetomidine in order to evaluate its efficacy in achieving pain control and comfort.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — administrating dexmedetomidine in order to evaluate the efficacy in achieving sedation for LISA procedure
  Other Names: LISA procedure

SUMMARY:
The investigators aim to evaluate: the effectiveness of dexmedetomidine for analgesia and sedation during LISA procedure, without compromising the respiratory drive; the safety of this drug on the preterm infant in a pilot study.

DETAILED DESCRIPTION:
Information will be given to parents of preterm babies <36 wGA upon their admission to the NICU (neonatal intensive care unit), and informed consent will be obtained as soon as possible. Eligible babies for LISA procedure (dyspneic and FiO2 > 0.30 on CPAP pressure of at least 6 cmH2O) undergo sedation with dexmedetomidine 1 mcg/kg, administered slowly iv in 10 minutes, together with non pharmacological techniques. After the step of sedation LISA is performed. Before/during and after the procedure pain will be assessed by the NIPS scale and the quality of intubation will be evaluated; then other events related to the procedure will be strictly collected for the first 24 hours. Babies will then be managed in usual NICU way and clinical data will be unregistered on respiratory, neurological and hemodynamic outcomes during the hospital stay, and especially at discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm newborns between 26+0 and 36+6 weeks of gestation stratified in two groups: VLBWI 26-31+6and LBWI 32-36+6.
2. Respiratory distress syndrome requiring surfactant therapy

Exclusion Criteria:

1. Need for emergency intubation in the delivery room
2. Major congenital malformations (such as cardiopathies)
3. Chromosomic abnormalities
4. Fetal Hydrops
5. Hypercapnia: CO2 > 65 mmHg
6. Pneumothorax
7. Hemodynamic compromise

Ages: 26 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
effectiveness of dexmedetomidine in achieving sedation for LISA procedure | basal (before procedure), during and immediately after the procedure
  evaluation of changes in Neonatal Infant Pain Scale (NIPS) score (0-2 points= no pain, 3-4 points = moderate pain; > 4 = severe pain)
Safety of dexmedetomidine in sedating preterm infants | 24 hours
  evaluation of number of apneas ( > 20 seconds or < 20 seconds with bradycardia < 100 bpm or desaturation ( SpO2 < 85%)); number of severe apnea and bradycardia (defined by the American Academy of Pediatrics Guidelines as apnea > 30 seconds and/or heart rate < 60 beats/minute for more than 10 seconds); need for intubation.

SECONDARY OUTCOMES:
number of laryngoscopies needed to perform LISA | during the procedure
  calculate the number of laryngoscopies needed to perform LISA
time needed to perform LISA | during the procedure
  calculate the time needed to perform LISA
Intubation conditions | during the procedure
  evaluated by the operator using the Goldberg scale (3 = excellent intubation conditions; 4-6= good intubation conditions; 7-9 = poor intubation conditions; 10-12 = inadequate intubation conditions)
the evolution of cardiorespiratory parameters | 1 min, 3 min, 5 min, 15 min, 30 min, 60 min and 120 min after the first drug injection
  heart rate (beats per minute)
the evolution of cardiorespiratory parameters | 1 min, 3 min, 5 min, 15 min, 30 min, 60 min and 120 min after the first drug injection
  respiratory rate (breaths per minute)
the evolution of cardiorespiratory parameters | 1 min, 3 min, 5 min, 15 min, 30 min, 60 min and 120 min after the first drug injection
  pulse oximetry (%)
the evolution of cardiorespiratory parameters | 1 min, 3 min, 5 min, 15 min, 30 min, 60 min and 120 min after the first drug injection
  blood pressure (mmHg)
the evolution of cardiorespiratory parameters | 1 min, 3 min, 5 min, 15 min, 30 min, 60 min and 120 min after the first drug injection
  FiO2 maxima during the procedure maintained for at least 30 seconds (%)
changes in ventilation mode | 1 min, 3 min, 5 min, 15 min, 30 min, 60 min and 120 min after the first drug injection
  inspiratory and end-expiratory ventilation pressures changes (cmH2O)
The incidence of drug adverse effects | 24 hours after drug injection
  respiratory events (i.e. bronchospasm) or cardiovascular events (bradycardia, hypotension)
The incidence of pneumothorax or selective administration of surfactant | 24 hours after drug injection
  RX evaluation
Long term outcomes | at 40 weeks PMA
  mortality (%)
Long term outcomes | at 40 weeks PMA
  bronchopulmonary dysplasia (%), defined as oxygen administration and/or respiratory support at 36 wGA
Long term outcomes | at 40 weeks PMA
  intraventricular hemorrhage (%) and periventricular leukomalacia (%)
Long term outcomes | at 40 weeks PMA
  necrotizing enterocolitis (%)
Long term outcomes | at 40 weeks PMA
  retinopathy of prematurity (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Paola Lago, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at the end of the study (April 2023)
Access Criteria: The investigators will access the data and the statistician

REFERENCES:
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Lemyre B, Laughon M, Bose C, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD005384. doi: 10.1002/14651858.CD005384.pub2. PMID 27976361
- [Background] Fischer HS, Buhrer C. Avoiding endotracheal ventilation to prevent bronchopulmonary dysplasia: a meta-analysis. Pediatrics. 2013 Nov;132(5):e1351-60. doi: 10.1542/peds.2013-1880. Epub 2013 Oct 21. PMID 24144716
- [Background] Jensen EA, DeMauro SB, Kornhauser M, Aghai ZH, Greenspan JS, Dysart KC. Effects of Multiple Ventilation Courses and Duration of Mechanical Ventilation on Respiratory Outcomes in Extremely Low-Birth-Weight Infants. JAMA Pediatr. 2015 Nov;169(11):1011-7. doi: 10.1001/jamapediatrics.2015.2401. PMID 26414549
- [Background] Verder H, Agertoft L, Albertsen P, Christensen NC, Curstedt T, Ebbesen F, Greisen G, Hobolth N, Holm V, Jacobsen T, et al. [Surfactant treatment of newborn infants with respiratory distress syndrome primarily treated with nasal continuous positive air pressure. A pilot study]. Ugeskr Laeger. 1992 Jul 27;154(31):2136-9. Danish. PMID 1509593
- [Background] Kribs A. Minimally Invasive Surfactant Therapy and Noninvasive Respiratory Support. Clin Perinatol. 2016 Dec;43(4):755-771. doi: 10.1016/j.clp.2016.07.010. Epub 2016 Oct 14. PMID 27837757
- [Background] Kribs A, Roll C, Gopel W, Wieg C, Groneck P, Laux R, Teig N, Hoehn T, Bohm W, Welzing L, Vochem M, Hoppenz M, Buhrer C, Mehler K, Stutzer H, Franklin J, Stohr A, Herting E, Roth B; NINSAPP Trial Investigators. Nonintubated Surfactant Application vs Conventional Therapy in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2015 Aug;169(8):723-30. doi: 10.1001/jamapediatrics.2015.0504. PMID 26053341
- [Background] Isayama T, Iwami H, McDonald S, Beyene J. Association of Noninvasive Ventilation Strategies With Mortality and Bronchopulmonary Dysplasia Among Preterm Infants: A Systematic Review and Meta-analysis. JAMA. 2016 Aug 9;316(6):611-24. doi: 10.1001/jama.2016.10708. PMID 27532916
- [Background] Aldana-Aguirre JC, Pinto M, Featherstone RM, Kumar M. Less invasive surfactant administration versus intubation for surfactant delivery in preterm infants with respiratory distress syndrome: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F17-F23. doi: 10.1136/archdischild-2015-310299. Epub 2016 Nov 15. PMID 27852668
- [Background] Kumar P, Denson SE, Mancuso TJ; Committee on Fetus and Newborn, Section on Anesthesiology and Pain Medicine. Premedication for nonemergency endotracheal intubation in the neonate. Pediatrics. 2010 Mar;125(3):608-15. doi: 10.1542/peds.2009-2863. Epub 2010 Feb 22. PMID 20176672
- [Background] COMMITTEE ON FETUS AND NEWBORN and SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE. Prevention and Management of Procedural Pain in the Neonate: An Update. Pediatrics. 2016 Feb;137(2):e20154271. doi: 10.1542/peds.2015-4271. Epub 2016 Jan 25. PMID 26810788
- [Background] Foglia EE, Ades A, Sawyer T, Glass KM, Singh N, Jung P, Quek BH, Johnston LC, Barry J, Zenge J, Moussa A, Kim JH, DeMeo SD, Napolitano N, Nadkarni V, Nishisaki A; NEAR4NEOS Investigators. Neonatal Intubation Practice and Outcomes: An International Registry Study. Pediatrics. 2019 Jan;143(1):e20180902. doi: 10.1542/peds.2018-0902. Epub 2018 Dec 11. PMID 30538147
- [Background] Descamps CS, Chevallier M, Ego A, Pin I, Epiard C, Debillon T. Propofol for sedation during less invasive surfactant administration in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2017 Sep;102(5):F465. doi: 10.1136/archdischild-2017-312791. Epub 2017 May 8. No abstract available. PMID 28483817
- [Background] Dekker J, Lopriore E, Rijken M, Rijntjes-Jacobs E, Smits-Wintjens V, Te Pas A. Sedation during Minimal Invasive Surfactant Therapy in Preterm Infants. Neonatology. 2016;109(4):308-13. doi: 10.1159/000443823. Epub 2016 Feb 24. PMID 26907795
- [Background] Bourgoin L, Caeymaex L, Decobert F, Jung C, Danan C, Durrmeyer X. Administering atropine and ketamine before less invasive surfactant administration resulted in low pain scores in a prospective study of premature neonates. Acta Paediatr. 2018 Jul;107(7):1184-1190. doi: 10.1111/apa.14317. Epub 2018 Apr 16. PMID 29532502
- [Background] Dekker J, Lopriore E, van Zanten HA, Tan RNGB, Hooper SB, Te Pas AB. Sedation during minimal invasive surfactant therapy: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F378-F383. doi: 10.1136/archdischild-2018-315015. Epub 2018 Aug 1. PMID 30068669
- [Background] Chevallier M, Durrmeyer X, Ego A, Debillon T; PROLISA Study Group. Propofol versus placebo (with rescue with ketamine) before less invasive surfactant administration: study protocol for a multicenter, double-blind, placebo controlled trial (PROLISA). BMC Pediatr. 2020 May 8;20(1):199. doi: 10.1186/s12887-020-02112-x. PMID 32384914
- [Background] Venkatraman R, Hungerford JL, Hall MW, Moore-Clingenpeel M, Tobias JD. Dexmedetomidine for Sedation During Noninvasive Ventilation in Pediatric Patients. Pediatr Crit Care Med. 2017 Sep;18(9):831-837. doi: 10.1097/PCC.0000000000001226. PMID 28598946
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] Tran DTT, Newton EK, Mount VAH, Lee JS, Mansour C, Wells GA, Perry JJ. Rocuronium vs. succinylcholine for rapid sequence intubation: a Cochrane systematic review. Anaesthesia. 2017 Jun;72(6):765-777. doi: 10.1111/anae.13903. PMID 28654173
- [Background] Eichenwald EC; Committee on Fetus and Newborn, American Academy of Pediatrics. Apnea of Prematurity. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3757. Epub 2015 Dec 1. PMID 26628729
- [Result] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433